CLINICAL TRIAL: NCT04435899
Title: Exercise Mediation on Hormonal, Immune and Psychological Well-being in Institutionalized Frail Older Women.
Acronym: UC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Guilherme Eustáquio Furtado, Researcher, principal investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University of Coimbra (CIDAF)
Record Dates: First submitted 2020-06-03; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Frail Elderly Syndrome
Keywords: Frail-older adults; disability; physical fitness; sex steroid hormones; cognition; motor skills
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EFFECTS OF A CHAIR-YOGA EXERCISES ON STRESS HORMONE LEVELS. (Experimental): assess the changes mediated by exercise on activities of daily life and falls (autonomy), physical fitness, salivary cortisol and alpha amylase in older adults living in social care givers centers. Methods: 35 women (83.81 ± 6.6 years old) were divided into two groups: chair-yoga exercises (CY, n=20) and control group (CG, n=15). All subjects were evaluated before and after 14-weeks of intervention. CY was involved in classes two times per week, while the GC did not participate in any exercise.
  Interventions: Other: Physical exercise
- Physical fralty and health outcomes of fitness, sex hormones. (Experimental): The study aimed to investigate the association of frailty with diverse geriatric health characteristics and how the latter might contribute to the former. Cross-sectional data of 140 women aged over 75 years were analyzed. Fried's definition of physical frailty, psychological, sex hormones, disability and physical fitness outcomes were examined. Prevalence of frailty was 40%. Frail women had lower scores in cognitive and physical fitness, and high scores for depression and comorbidities. Significant correlations emerged between frailty and disability, fear of falling, aerobic resistance and cognition showed that only aerobic resistance and cognition. A trend towards lower systolic blood pressure in the frail group may reflect being less physically active and/or having more systemic comorbidity. Using simple functional fitness and cognitive measures rather than using less reliable self-report assessments can better identify those with physical frailty.
  Interventions: Other: Physical exercise
- physical fitness and frailty syndrome institutionalized older (Experimental): This study analyzed the relationship between old physical frailty syndrome (PF) and PhFi indicators and assessed how the latter might predict the former. Participants were 119 elderly women (81.96 ±7.89 years) recruited from four social and healthcare centers. PhFi was assessed through muscle strength tests of upper and lower limbs, endurance, agility-dynamic balance, flexibility and body composition.
  The following PF indicators were assessed: weight loss, exhaustion, weakness, slowness and low physical activity level.
  Interventions: Other: Physical exercise
- THE RELATIONSHIP BETWEEN FUNCTIONAL DISABILITY OUTCOMES (Experimental): The associations between functional disability activities of life activities and frailty have already been explored. The contribution of each component of physical frailty and their contribution to understanding the early physical decline of older individuals are poorly explored. The relationships between PF and functional disability and to identify the independent components of frailty that most influence on disability in older women. A cross-sectional study of 119 (81,96±7,89) older women aged 75 and over. Functional disability was assessed through Agility-dynamic and Static balance tests, Activities of daily life and Falls risk screen outcomes.
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: Physical exercise — Multi-modal exercise protocol

SUMMARY:
Frailty syndrome is a complex aging expression determined by ontogenetic and phylogenetic factors. Chronic stress has been shown to have immunosuppressive effects, to accelerate immunosenescence and to cause cumulative disorders in many physiological systems, resulting in frail state. In a recent approach, Linda Fried and colleagues have developed a construct whose bases are muscle loss, negative energy balance and physical inactivity, called 'Frailty Cycle'. They identified five dimensions in the construct: weakness, low resistance to an effort, slowness, low physical activity, and weight loss, which were operationalized on five criteria to identify the Physical Frailty (PF), and divide the population in frail, pre-frail and non-frail. Recently, epidemiological studies reported that cognitive impairments, low immune expression, and others global health dimensions have a powerful association with physical frailty. However, there is a need for the search for new correlated markers for the frail condition, for a better understanding of the phenomenon. On the other hand, exercise has been shown as a co-adjuvant treatment to have positive effects on several factors linked to physical frailty (e.g. improve immunity and prevent chronic diseases), because of it's potential effect on hormonal mediation. Looking at Fried PF Phenotype construct, their dimensions share biological 'commonalities' that can be explained by studying the biopsychological mechanisms with exercise being a key factor in the study of these relationships.

The current research was designed to investigate and characterize the prevalence of the PF in a cross-sectional Portuguese samples (institutionalized participants), to examine the relationship between PF and each one of the general health status domain such as physical fitness and functioning status; neuroendocrine and immune parameters; psychological and cognitive ability of these populations; and to verified the impact of different types of exercise in each domain of general health status. However, this doctoral thesis is presented in the form of articles, divided into five sections and their respective chapters. In total, 3 preliminary studies (2 systematic reviews of studies 1 and 2 and one exercise-intervention pilot study 3), 5 cross-sectional studies (4,5,6,7, and 8) and 3 intervention studies (9,10 and 11) were completed. The cross-sectional design consisted of the assessment of 140 older women (≥75 years old), living in different centres of heath care and social support, located in the city of Coimbra, Portugal. The participants were selected using a non-probabilistic convenience sampling based on the geographical area of the center region of Coimbra city.

DETAILED DESCRIPTION:
This research protocol was planned for approximately 13 months, involving a trained research team and it is built in different phases, according to the type of studies: cross- sectional and experimental. The cross-sectional study (4 weeks' duration) consisted in the evaluation of older people (65 years old), living in different centres of heath care and social support (HCS), located in the city of Coimbra, Portugal. The participants were selected using a non-probalistic convenience sampling based on the geographical area of center region of Coimbra city. The experimental phase characterized as an intervention study with two different chair-based exercise programs, designed to assess the effect of strength/elastic band and multimodal interventions on biopsychological outcomes in frail e pre- frail individuals. Participants in these groups was attended a 45 minutes' exercise session, two-three times per week during 28 weeks and were extracted using the Physical Frailty status from the cross-sectional study design.

ELIGIBILITY:
Inclusion Criteria:

* inclusion criteria: a) ability to participate in a study with total duration of 12 months and encompassing three phases: cross-sectional study, intervention and detraining periods b) existence of an appropriate physical space to carry out the exercise sessions; c) required support of caregivers to assist with the elders' displacement to the exercise classes;

Exclusion Criteria:

* The following selection criteria for participants included was adopted: a) take a part in this study spontaneously; b) drug therapy and clinical condition controlled and updated (it must be stable and enable participation in the exercise classes as decided by local medical staff); c) not completing the '8-foot-up and go test' in the maximum time of 50 seconds.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
physical exercise | 14 weeks
  weight and height will be combined to report BMI in kg/m2

CONTACTS AND LOCATIONS:
Locations (1):
- Care Centers, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Undecided